CLINICAL TRIAL: NCT03308643
Title: Effect of Oxytocin Infusion on Blood Loss During Abdominal Myomectomy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Kanuni Sultan Suleyman Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Berna Aslan Cetin, Attending physician,ObGyn, Kanuni Sultan Suleyman Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2016/3
Record Dates: First submitted 2017-10-09; First posted 2017-10-12 (Actual); Last update posted 2018-05-21 (Actual); Status verified 2018-05

CONDITIONS: Myomectomy
Keywords: myomectomy; oxytocin; blood loss
MeSH Terms: conditions — Hemorrhage | interventions — Oxytocin; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: The abdominal myomectomy cases will be randomized into 2 separate groups in a parallel fashion using an online software at 1:1 ratio.
Who Masked: Participant, Investigator
Masking Description: Randomization will be performed by an online software and the list will be given to anesthesiologist so that neither the surgeon nor patient will know which intervention was performed. Randomized cards will be in sealed envelopes and will be open by anesthesiologist at the time of surgery.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oxytocin infusion (Experimental): Patients will receive intravenous oxytocin infusion just before the surgery after the induction of general anesthesia.
  Interventions: Drug: Oxytocin
- Placebo (Placebo Comparator): Patients will receive pure normal saline infusion at the same rate and volume just before the surgery after the induction of general anesthesia.
  Interventions: Other: saline

INTERVENTIONS:
Drug: Oxytocin — Patients will receive intravenous oxytocin infusion just before the surgery after the induction of general anesthesia.
  Arms: Oxytocin infusion
Other: saline — Patients will receive intravenous normal saline infusion just before the surgery after the induction of general anesthesia.
  Arms: Placebo

SUMMARY:
To evaluate the effects of oxytocin infusion during abdominal myomectomy.

DETAILED DESCRIPTION:
Myomectomy is indicated for symptomatic uterine fibroids. Fibroids have blood supply and 20% of the abdominal myomectomy cases might require blood transfusion because of the nature of the surgery. Oxytocin infusion is one of the intervention to decrease blood loss during myomectomy. To evaluate the effects and benefits of oxytocin infusion during abdominal myomectomy we decide to conduct this randomized study.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-50
* Patients who are candidate for abdominal myomectomy

Exclusion Criteria:

* History of previous myomectomy.
* Suspected malignancy
* Patients with preoperative anemia
* Patients using hormonal treatments before the surgery.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Female patients with uterus and undergoing abdominal myomectomy
Enrollment: 100 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2018-05-10 (Actual); Study Completion 2018-05-10 (Actual)

PRIMARY OUTCOMES:
Blood loss during surgery | 2 hours
  estimated blood loss during the surgery measured by aspiration fluid.

SECONDARY OUTCOMES:
Blood loss after abdominal myomectomy | 1 hour postoperatively
  change in Hematocrit Percentage (before and after the surgery)

CONTACTS AND LOCATIONS:
Overall Officials: Berna Aslan, Study Director — Kanuni Sultan Suleyman Research and Training Hospital
Locations (1):
- Kanuni Sultan Suleyman Egitim ve Arastırma Hastanesi, Istanbul, Turkey (Türkiye)

REFERENCES:
- [Result] Atashkhoei S, Fakhari S, Pourfathi H, Bilehjani E, Garabaghi PM, Asiaei A. Effect of oxytocin infusion on reducing the blood loss during abdominal myomectomy: a double-blind randomised controlled trial. BJOG. 2017 Jan;124(2):292-298. doi: 10.1111/1471-0528.14416. Epub 2016 Nov 15. PMID 27862855
- [Result] Chang FW, Yu MH, Ku CH, Chen CH, Wu GJ, Liu JY. Effect of uterotonics on intra-operative blood loss during laparoscopy-assisted vaginal hysterectomy: a randomised controlled trial. BJOG. 2006 Jan;113(1):47-52. doi: 10.1111/j.1471-0528.2005.00804.x. PMID 16398771